CLINICAL TRIAL: NCT02672189
Title: A Randomized Controlled Trial of Internet-based Cognitive Behavioral Therapy for Breast Cancer Patients With Climacteric Symptoms
Brief Title: Internet-based Cognitive Behavioral Therapy for Breast Cancer Patients With Climacteric Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKI 2014-6788 / NL53182.031.15
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Climacteric Symptoms; Breast Cancer Survivors
Keywords: Climacteric symptoms; Menopause; Breast Cancer Survivors; Internet-based; Cognitive behavioral therapy; Psychosocial intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waiting list control group (No Intervention): Women in the waiting list control group will receive usual care. They will complete questionnaires during a period of 6 months. After completion of the last questionnaire they will be offered the opportunity to follow the EVA-Online program.
- EVA-Online guided group (Experimental): The CBT/Relaxation program (EVA-Online) consists of 6 online sessions intended to be completed weekly over a 6 week period. The program comprises the following elements: (1) information and advice about symptoms (e.g., hot flushes, night sweats and sexual functioning); (2) monitoring and modifying precipitants; (3) relaxation and stress reduction; (4) cognitive restructuring of unhelpful thoughts and (5) encouraging helpful behavioral strategies (e.g., pacing activities). Throughout the program women will be asked to spend an hour a week to read the session and fill in the assignments and to spend 30 minutes per day on homework exercises (eg, filling in a hot flush/night sweats diary, practicing relaxation techniques).
  Participating women will first undergo a 30 minute phone interview with a trained therapist before they start the online program. The same therapist will provide weekly feedback and support.
  Interventions: Behavioral: EVA-Online
- EVA-Online self-management group (Experimental): The content of the self-management CBT/Relaxation program is the same as the guided version of the program as described above, but without weekly guidance by a trained therapist. The women allocated to the self-management intervention will work through the program independently.
  Interventions: Behavioral: EVA-Online

INTERVENTIONS:
Behavioral: EVA-Online — Internet-based cognitive behavioral therapy
  Arms: EVA-Online guided group; EVA-Online self-management group

SUMMARY:
The current study will evaluate systematically the efficacy and cost-effectiveness of two internet-based CBT/relaxation programs (one guided, the other self-managed) in reducing the severity of menopausal symptoms and improving copings skills with regard to hot flushes and night sweats as well as improving sexual functioning, improving quality of sleep, reducing emotional distress and improving quality of life in younger breast cancer patients who experience treatment-induced menopause.

DETAILED DESCRIPTION:
Background: Breast cancer is the most common cancer among women in the Netherlands, with approximately 14.000 new cases reported in 2011 (1). Nearly 30% of all women with breast cancer are premenopausal at the time of diagnosis (2). Ovarian damage is a major long-term sequela of chemotherapy in premenopausal women (3,4). Ovarian failure induced by chemotherapy and/or endocrine treatment leads to an earlier onset of menopause, with age and duration of treatment being its strongest predictors (5).

Premature menopause is a major concern of younger women undergoing (adjuvant/preventive) therapy for cancer (6). Primary menopausal symptoms include hot flushes, night sweats, vaginal dryness, decreased libido, dysuria and urinary incontinence. Secondary symptoms include insomnia due to night sweats, dyspareunia because of vaginal dryness, weight gain, and psychological distress (3,7,8). Previous studies have indicated that the severity of hot flushes is increased in women who experience transition into menopause during cancer treatment or after PBSO, compared to women going through natural menopause (9,10,11).

Among menopausal symptoms, hot flushes are considered to be the most disruptive, with prevalence rates between 63% and 80% in breast cancer patients (7,12-15). Moreover, vasomotor symptoms are an important reason why some women discontinue tamoxifen treatment (16,17). Hormonal replacement therapy (HRT) is highly effective in alleviating vasomotor symptoms associated with menopause (18). However, HRT is contraindicated in women with a history of breast cancer (19), even after prophylactic bilateral salpingo oophorectomy (PBSO) (20).

There is increasing evidence that behavioral interventions have a positive impact on symptoms in women with naturally occurring and treatment-induced menopause (21-27). A cognitive behavioral therapy (CBT) intervention including information about symptoms, monitoring and modifying precipitants, relaxation and stress management, cognitive restructuring of unhelpful assumptions and automatic thoughts, and encouraging helpful behavioral strategies has been found to be beneficial in the alleviation of menopausal symptoms in women with breast cancer (25,26), but compliance with face-to-face CBT programs can be problematic (26). A promising approach is to make this form of CBT more accessible and feasible for participants by having it available via the internet. Although the efficacy of CBT for this patient population has been demonstrated in the form of face-to-face group therapy, its efficacy has not been investigated when delivered via an internet platform in an individual setting.

Design. For this trial patients will be recruited from several hospitals in the Netherlands (predominantly Amsterdam region). Participants will be randomly allocated to either the guided intervention group, the self-management group or the control group (N = 83 per group). Upon completion of the study, the patients assigned to the control group will be given the opportunity to undergo the internet-based cognitive behavioral therapy program.

Women in the two intervention and control group will be asked to complete a battery of questionnaires prior to randomization (TO), at 10 weeks (T1) and at 6 months (T2).

Study measures. The primary outcomes are menopausal complaints, as assessed with a menopausal complaints questionnaire, the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES), and hot flushes and night sweats as assessed by the Hot Flushes Rating Scale (HFRS). The secondary study outcomes are sexuality problems (the Sexual Activity Questionnaire (SAQ)); sleep quality (The Groningen Sleep Quality Score (GSQS)); psychological distress (The Hospital Anxiety and Depression Scale (HADS)) and health related quality of life (The Medical Outcome Study 36-Item Short Form-36 Health Survey (SF-36)).

Patients' evaluation of the intervention program. The women in both intervention groups will be asked to provide their opinion of the internet-based CBT program at the 10 week evaluation point. All these women will be asked to complete a short questionnaire about the perceived efficacy of and satisfaction with the intervention program, whether they would suggest any changes to the program, and if they would recommend it to other women experiencing symptoms of premature menopause. In addition, telephone interviews (30 minutes) will be held with women who: (1) stated in the questionnaire that the intervention did not have the desired effect; and/or (2) gave the intervention a low rating (<6) and/or (3) would not recommend the program to others.

Cost effectiveness. The cost-effectiveness of the internet-based guided CBT versus the internet-based self-management CBT versus usual care will be expressed as: (1) cost per patient with a clinically relevant significant reduction on the HFRS and (2) cost per quality adjusted life year (QALY) gained.

Sample size and statistical power calculations: In total, 248 women will be recruited into the study, to allow for an attrition rate of approximately 20% (i.e., women who discontinue participation in the study entirely, including failure to complete all follow-up questionnaires; those women who discontinue participation in one of the groups but complete the follow-up assessments will be included in the analysis). Thus, a minimum of 130 women will be available for the primary intention-to-treat analysis. With a total sample of 130 women (65 per group), the study will have 80% power to detect an effect size of 0.5 with a p value of 0.05 (28).

Statistical analyses: Analyses will first be performed to evaluate the comparability of the intervention groups (guided versus self-management) and control group at baseline in terms of sociodemographic and clinical characteristics. ANOVA tests or appropriate non-parametric statistics will be used, depending on the level of measurement. If, despite the stratified randomization procedures, the groups are found not to be comparable on one more background variables, those variables will be employed routinely as covariates in subsequent analyses.

We will evaluate between-group differences over time in self-reported endocrine symptoms, sexual functioning, psychological distress, sleep quality and HRQOL. Scores for the FACT-ES, the HFRS, the SAQ, the HADS, the GSQS, and the SF-36 and the utility version of the SF-36, the SF-6D will be calculated according to published scoring algorithms.We will compare both intervention groups with the control group over time using multilevel procedures with repeated measures, using a restricted maximum likelihood (REML) solution to model specific contrasts between groups and follow-up assessment (29). Within each multilevel model the control group will be the reference category. Differences in mean change scores over time between the intervention groups and the control group will be accompanied by effect sizes (ES). As indicated previously, the FACT-ES and the HFRS will be used as the primary study endpoints, and the remaining measures will be considered as secondary endpoints. The p-value for overall model effects will be set at 0.05, and for specific contrasts at 0.01, lowering the risk of Type errors due to multiple testing.

All analyses will be conducted on an intention-to-treat (ITT) basis. In addition, per-protocol (PP) analyses will be performed on patients who met criteria for minimal compliance with the intervention(s). Supplementary analyses will be carried out in which data relating to compliance with the program elements is taken into account. Specifically, we will determine whether the level of compliance (based on completed homework assignments and self-report data) is associated significantly with the changes over time in symptom relief, sexuality, psychological distress, sleep quality, and cost-effectiveness. In addition the potential mediating effect of hot flush beliefs and behaviors will be examined through mediator analysis.

A cost-effectiveness analysis (CEA) will be performed using a validated health economic model as developed for use in the EVA-Trial (30). The analysis will consider the societal perspectives, the third-party payer perspective and the healthcare system perspective in comparing the effectiveness and costs of web-based CBT for alleviating treatment-induced menopausal symptoms versus waiting list control. Effectiveness data as gathered from the trial will be combined with the cost data from the cost-diary and hospital administration data.

ELIGIBILITY:
Age limit: stated age concerns age at time of diagnosis.

Inclusion Criteria:

* Female
* Diagnosis of histologically confirmed primary breast cancer
* 50 years or younger at time of diagnosis
* Premenopausal at time of diagnosis
* Treatment induced menopause due to at least one of the following treatment regimens: 1) chemotherapy (< 5 years > 4 months); 2) hormonal therapy (<5 years; may currently receive hormonal treatment); oophorectomy (< 5 years > 4 months)
* Disease free at time of study entry
* Presence of menopausal symptoms

Exclusion Criteria:

* Lacks basic proficiency in Dutch
* No access to the internet
* Serious cognitive or psychiatric problems
* Participation in concurrent studies and/or therapy programs to alleviate menopausal symptoms

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in overall levels of menopausal symptoms | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Overall levels of menopausal symptoms are assessed by using the FACT-ES
Change in vasomotor symptoms | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Vasomotor symptoms are assessed with the Hot Flush Rating Scale (HFRS)

SECONDARY OUTCOMES:
Change in overall levels of sexual functioning | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  The overall levels of sexual functioning are assessed with the Sexual Activity Questionnaire (SAQ)
Change in psychological distress | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Psychological distress is assessed with the Hospital Anxiety and Depression Scale (HADS)
Change in sleep quality | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Sleep quality is assessed with the Groningen Sleep Quality Scale (GSQS)
Change in hot flush frequency | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Hot flush frequency is assessed with the frequency subscale of the Hot Flush Rating Scale (HFRS)
Change in health related quality of life | Baseline (T0); 10 weeks post baseline (T1) and 6 months post baseline (T2)
  Health related quality of life is assessed with the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neil K. Aaronson, PhD, Principal Investigator — The Netherlands Cancer Institute; Hester S.A. Oldenburg, PhD, Principal Investigator — The Netherlands Cancer Institute; Marc Van Beurden, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Background] Cijfers over kanker, Nederlandse Kankerregistratie,beheerd door IKNL © januari 2014, 2014
- [Background] Society. AC: Cancer Facts Figures - 2000. Atlanta, GA, 2003
- [Background] Bines J, Oleske DM, Cobleigh MA. Ovarian function in premenopausal women treated with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1996 May;14(5):1718-29. doi: 10.1200/JCO.1996.14.5.1718. PMID 8622093
- [Background] Shapiro CL, Recht A. Side effects of adjuvant treatment of breast cancer. N Engl J Med. 2001 Jun 28;344(26):1997-2008. doi: 10.1056/NEJM200106283442607. No abstract available. PMID 11430330
- [Background] Goodwin PJ, Ennis M, Pritchard KI, Trudeau M, Hood N. Risk of menopause during the first year after breast cancer diagnosis. J Clin Oncol. 1999 Aug;17(8):2365-70. doi: 10.1200/JCO.1999.17.8.2365. PMID 10561298
- [Background] Avis NE, Crawford S, Manuel J. Psychosocial problems among younger women with breast cancer. Psychooncology. 2004 May;13(5):295-308. doi: 10.1002/pon.744. PMID 15133771
- [Background] Couzi RJ, Helzlsouer KJ, Fetting JH. Prevalence of menopausal symptoms among women with a history of breast cancer and attitudes toward estrogen replacement therapy. J Clin Oncol. 1995 Nov;13(11):2737-44. doi: 10.1200/JCO.1995.13.11.2737. PMID 7595732
- [Background] Biglia N, Cozzarella M, Cacciari F, Ponzone R, Roagna R, Maggiorotto F, Sismondi P. Menopause after breast cancer: a survey on breast cancer survivors. Maturitas. 2003 May 30;45(1):29-38. doi: 10.1016/s0378-5122(03)00087-2. PMID 12753941
- [Background] Rosenberg SM, Partridge AH. Premature menopause in young breast cancer: effects on quality of life and treatment interventions. J Thorac Dis. 2013 Jun;5 Suppl 1(Suppl 1):S55-61. doi: 10.3978/j.issn.2072-1439.2013.06.20. PMID 23819028
- [Background] Crandall C, Petersen L, Ganz PA, Greendale GA. Association of breast cancer and its therapy with menopause-related symptoms. Menopause. 2004 Sep-Oct;11(5):519-30. doi: 10.1097/01.gme.0000117061.40493.ab. PMID 15356404
- [Background] Benshushan A, Rojansky N, Chaviv M, Arbel-Alon S, Benmeir A, Imbar T, Brzezinski A. Climacteric symptoms in women undergoing risk-reducing bilateral salpingo-oophorectomy. Climacteric. 2009 Oct;12(5):404-9. doi: 10.1080/13697130902780846. PMID 19479488
- [Background] Bloom JR, Stewart SL, Chang S, Banks PJ. Then and now: quality of life of young breast cancer survivors. Psychooncology. 2004 Mar;13(3):147-60. doi: 10.1002/pon.794. PMID 15022150
- [Background] Carpenter JS, Andrykowski MA, Cordova M, Cunningham L, Studts J, McGrath P, Kenady D, Sloan D, Munn R. Hot flashes in postmenopausal women treated for breast carcinoma: prevalence, severity, correlates, management, and relation to quality of life. Cancer. 1998 May 1;82(9):1682-91. PMID 9576289
- [Background] Carpenter JS, Andrykowski MA. Menopausal symptoms in breast cancer survivors. Oncol Nurs Forum. 1999 Sep;26(8):1311-7. PMID 10497770
- [Background] Hunter MS, Grunfeld EA, Mittal S, Sikka P, Ramirez AJ, Fentiman I, Hamed H. Menopausal symptoms in women with breast cancer: prevalence and treatment preferences. Psychooncology. 2004 Nov;13(11):769-78. doi: 10.1002/pon.793. PMID 15386641
- [Background] Owusu C, Buist DS, Field TS, Lash TL, Thwin SS, Geiger AM, Quinn VP, Frost F, Prout M, Yood MU, Wei F, Silliman RA. Predictors of tamoxifen discontinuation among older women with estrogen receptor-positive breast cancer. J Clin Oncol. 2008 Feb 1;26(4):549-55. doi: 10.1200/JCO.2006.10.1022. Epub 2007 Dec 10. PMID 18071188
- [Background] Lash TL, Fox MP, Westrup JL, Fink AK, Silliman RA. Adherence to tamoxifen over the five-year course. Breast Cancer Res Treat. 2006 Sep;99(2):215-20. doi: 10.1007/s10549-006-9193-0. Epub 2006 Mar 16. PMID 16541307
- [Background] MacLennan A, Lester S, Moore V. Oral oestrogen replacement therapy versus placebo for hot flushes. Cochrane Database Syst Rev. 2001;(1):CD002978. doi: 10.1002/14651858.CD002978. PMID 11279791
- [Background] Holmberg L, Anderson H; HABITS steering and data monitoring committees. HABITS (hormonal replacement therapy after breast cancer--is it safe?), a randomised comparison: trial stopped. Lancet. 2004 Feb 7;363(9407):453-5. doi: 10.1016/S0140-6736(04)15493-7. PMID 14962527
- [Background] Finch A, Evans G, Narod SA. BRCA carriers, prophylactic salpingo-oophorectomy and menopause: clinical management considerations and recommendations. Womens Health (Lond). 2012 Sep;8(5):543-55. doi: 10.2217/whe.12.41. PMID 22934728
- [Background] Hunter MS: Cognitive behavioural interventions for premenstrual and menopausal problems. J Reprod Infant Psychol:183-193, 2003
- [Background] Irvin JH, Domar AD, Clark C, Zuttermeister PC, Friedman R. The effects of relaxation response training on menopausal symptoms. J Psychosom Obstet Gynaecol. 1996 Dec;17(4):202-7. doi: 10.3109/01674829609025684. PMID 8997686
- [Background] Lindh-Astrand L, Nedstrand E, Wyon Y, Hammar M. Vasomotor symptoms and quality of life in previously sedentary postmenopausal women randomised to physical activity or estrogen therapy. Maturitas. 2004 Jun 15;48(2):97-105. doi: 10.1016/S0378-5122(03)00187-7. PMID 15172083
- [Background] Ayers B, Smith M, Hellier J, Mann E, Hunter MS. Effectiveness of group and self-help cognitive behavior therapy in reducing problematic menopausal hot flushes and night sweats (MENOS 2): a randomized controlled trial. Menopause. 2012 Jul;19(7):749-59. doi: 10.1097/gme.0b013e31823fe835. PMID 22336748
- [Background] Mann E, Smith MJ, Hellier J, Balabanovic JA, Hamed H, Grunfeld EA, Hunter MS. Cognitive behavioural treatment for women who have menopausal symptoms after breast cancer treatment (MENOS 1): a randomised controlled trial. Lancet Oncol. 2012 Mar;13(3):309-18. doi: 10.1016/S1470-2045(11)70364-3. Epub 2012 Feb 15. PMID 22340966
- [Background] Duijts SF, van Beurden M, Oldenburg HS, Hunter MS, Kieffer JM, Stuiver MM, Gerritsma MA, Menke-Pluymers MB, Plaisier PW, Rijna H, Lopes Cardozo AM, Timmers G, van der Meij S, van der Veen H, Bijker N, de Widt-Levert LM, Geenen MM, Heuff G, van Dulken EJ, Boven E, Aaronson NK. Efficacy of cognitive behavioral therapy and physical exercise in alleviating treatment-induced menopausal symptoms in patients with breast cancer: results of a randomized, controlled, multicenter trial. J Clin Oncol. 2012 Nov 20;30(33):4124-33. doi: 10.1200/JCO.2012.41.8525. Epub 2012 Oct 8. PMID 23045575
- [Background] Ganz PA, Greendale GA, Petersen L, Zibecchi L, Kahn B, Belin TR. Managing menopausal symptoms in breast cancer survivors: results of a randomized controlled trial. J Natl Cancer Inst. 2000 Jul 5;92(13):1054-64. doi: 10.1093/jnci/92.13.1054. PMID 10880548
- [Background] Cohen J: Statistical power analysis for the behavioral sciences. Hillsdale, New Jersey, Lawrence Earlbaum Associates, 1988
- [Background] Diggle P, Heagerty P, Liang K, et al: Analysis of longitudinal data. New York, Oxford University Press, 2002
- [Background] Mewes JC, Steuten LM, Duijts SF, Oldenburg HS, van Beurden M, Stuiver MM, Hunter MS, Kieffer JM, van Harten WH, Aaronson NK. Cost-effectiveness of cognitive behavioral therapy and physical exercise for alleviating treatment-induced menopausal symptoms in breast cancer patients. J Cancer Surviv. 2015 Mar;9(1):126-35. doi: 10.1007/s11764-014-0396-9. Epub 2014 Sep 2. PMID 25179578
- [Derived] Atema V, van Leeuwen M, Kieffer JM, Oldenburg HSA, van Beurden M, Hunter MS, Aaronson NK. Internet-based cognitive behavioral therapy aimed at alleviating treatment-induced menopausal symptoms in breast cancer survivors: Moderators and mediators of treatment effects. Maturitas. 2020 Jan;131:8-13. doi: 10.1016/j.maturitas.2019.09.007. Epub 2019 Sep 18. PMID 31787152
- [Derived] Atema V, van Leeuwen M, Kieffer JM, Oldenburg HSA, van Beurden M, Gerritsma MA, Kuenen MA, Plaisier PW, Lopes Cardozo AMF, van Riet YEA, Heuff G, Rijna H, van der Meij S, Noorda EM, Timmers GJ, Vrouenraets BC, Bollen M, van der Veen H, Bijker N, Hunter MS, Aaronson NK. Efficacy of Internet-Based Cognitive Behavioral Therapy for Treatment-Induced Menopausal Symptoms in Breast Cancer Survivors: Results of a Randomized Controlled Trial. J Clin Oncol. 2019 Apr 1;37(10):809-822. doi: 10.1200/JCO.18.00655. Epub 2019 Feb 14. PMID 30763176
- [Derived] Atema V, van Leeuwen M, Oldenburg HS, Retel V, van Beurden M, Hunter MS, Aaronson NK. Design of a randomized controlled trial of Internet-based cognitive behavioral therapy for treatment-induced menopausal symptoms in breast cancer survivors. BMC Cancer. 2016 Nov 25;16(1):920. doi: 10.1186/s12885-016-2946-1. PMID 27887581